CLINICAL TRIAL: NCT01598701
Title: The Opioid-Sparing and Analgesic Effects of IV Acetaminophen in Craniotomy: A Prospective, Randomized, Placebo-Controlled, Double-Blind Study
Brief Title: Intravenous Acetaminophen in Craniotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Carlos Artime, Assistant Professor - Anesthesiology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HSC-MS-12-0055
Record Dates: First submitted 2012-05-09; First posted 2012-05-15 (Estimated); Results first posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Postoperative Pain
Keywords: Acetaminophen; Intravenous Acetaminophen; Opioid Requirement; Pain; Post-Operative Pain; Craniotomy; Post-Craniotomy Pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Acetaminophen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Acetaminophen (Experimental): Patients will be receive doses of 1000 mg/100 mL of IV Acetaminophen (OFIRMEV). The drug will be infused over 15 minutes.
  Interventions: Drug: Acetaminophen
- Placebo (Placebo Comparator): Patients will be given 100 mL normal saline placebos at scheduled time intervals in place of IV acetaminophen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetaminophen — Intravenous Acetaminophen, 1000 mg/100mL, Every 6 hours, Infused over 15 minutes.
  Other Names: OFIRMEV
  Arms: Intravenous Acetaminophen
Drug: Placebo — 100 mL 0.9% Sodium Chloride
  Other Names: 0.9% Sodium Chloride
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the use of intravenous Acetaminophen (OFIRMEV) as an effective adjunct therapeutic agent in patients undergoing craniotomy.

DETAILED DESCRIPTION:
General anesthesia will be induced by bolus administration of propofol (1.5-2.5 mg/kg IV), and fentanyl (2-3 µg/kg IV). Neuromuscular blockade will be achieved with bolus administration of rocuronium, vecuronium, or succinylcholine. Once the endotracheal tube is secured in place, the patient will be mechanically ventilated to an end-tidal CO2 of 35 mmHg. Additional procedures will include radial arterial line placement for invasive arterial blood pressure monitoring, as well as additional large-bore peripheral IV placements, or central line placement, if indicated. Anesthesia will be maintained with desflurane, propofol, and remifentanil.

Once general anesthesia has been induced, but prior to the first surgical incision, the first dose of the interventional agent will be administered. Repeat doses will be administered every 6 hours until 24 hours from the time that the patient enters the PACU, for a total of up to 6 doses. Once the patient has been positioned and prepped for surgery, the surgeon will infiltrate the scalp with bupivacaine 0.5% with epinephrine 1:200,000 (15-20 ml) before skin incision.

No other opioids or agents with analgesic properties (e.g., ketorolac, dexmedetomidine, ketamine) will be administered at any time during the operation. Additional medications that will be routinely administered for this procedure include dexamethasone 8-12mg IV prior to incision, and ondansetron 4mg IV at skin closure. Anticonvulsant drugs will be administered at the surgeon's request.

Emergence and extubation will occur at the completion of the case per standard guidelines. The time of remifentanil infusion discontinuation and time of extubation will be noted. If necessary, extubation may occur in the post anesthesia recovery unit (PACU); otherwise, extubation will occur in the operating room.

The patient will then be taken directly to the PACU. Inability to extubate a patient within two hours of completion of surgery will result in their withdrawal from the study. Once in the PACU, immediate postoperative vital signs will be recorded, including blood pressure, heart rate, respiratory rate, oxygen saturation, and RASS score.

Pain scores will be assessed using the visual analog scale (VAS) upon entering the PACU or upon extubation in PACU (0 hours), and then again at 1, 2, 4, 8, 12, 16, 20, and 24 hours post-operatively. The VAS will be a 10 cm scale on a numerical scale of 0 (no pain) to 10 (severe pain) that the patient will point to in order to indicate their current level of pain. Pain scores will be measured while the patient is at rest. Post-operative nausea will also be recorded on a 10 cm numeric rating scale (NRS) at the same time intervals, with 0 indicating no nausea and 10 indicating severe nausea. All day-time VAS and NRS measurements will be made by a research assistant. Night-time measurements will be made by the nurse on the unit.

While in the PACU, the time until the patient receives their first dose of analgesic medicine will be recorded. Patients will be given a 2mg nurse-administered dose of morphine upon request or if they report a pain score of ≥4/10, and will continue to be given morphine doses based on clinical assessment by the PACU/intensive care nurse, who will be blind to patient group allocation. The nurse will objectively assess the patient's pain score at least once an hour using the VAS pain scale, and an assessment of pain ≥4/10 will warrant an additional 2mg dose of morphine. Morphine dosage requirements will be recorded for 24 hours post-operatively. If morphine requirement is greater than 10mg in a 30 minute period or the patient develops an allergic reaction, pruritus, renal insufficiency, drowsiness, nausea/vomiting, or clinically relevant reason to change medication, the PACU supervising physician or ICU physician may use their clinical discretion to change the opioid rescue medication to hydromorphone (0.3mg doses). The reason for changing medication will be reported by the physician and recorded. The morphine equivalent of hydromorphone will be estimated to be 7 times the hydromorphone dose. The PACU/ICU nurses will also record any episodes of emesis, use of rescue anti-emetic medicine, and the occurrence of any other side effects.

A post-operative neurologic examination will take place in the PACU. Criteria for a neurological exam to be complete is the patient's ability to successfully lift each leg off of the bed for more than two seconds on command, and to be able to hold up two fingers on each hand on command. If these criteria are not met prior to transferring the patient from the PACU to the ICU, a post-operative neurologic complication will be considered and the patient will be withdrawn from the study.

The time until the patient is ready to be discharged from the PACU will also be noted. Patients with a modified Aldrete score of ≥ 8 (see Appendix 1) will be considered ready for discharge. These criteria will be assessed by either the research assistant or PACU staff.

At the end of the 24 hour post-operative time period, a patient interview will be conducted. At this interview the patient will asked about their subjective satisfaction with their analgesic protocol, as well as any adverse effects they may have noticed. The 24 hour morphine consumption will also be recorded at this time.

After the study is completed, patients may receive IV or oral acetaminophen therapy at the discretion of the primary physician.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Undergoing Craniotomy for Supratentorial Tumor Resection
* Weight between 50 and 120 kilograms
* ASA Physical Status I-III
* Be able to communicate verbally
* Be able to use Visual Analog Score

Exclusion Criteria:

* Allergies to acetaminophen, morphine or any of the anesthetic agents required by the protocol.
* Use of opioids, tramadol, benzodiazepines, or gabapentin on a daily basis for > 7 days prior to the day of surgery.
* Use of acetaminophen, NSAIDs, or any other analgesic medication in the 12 hours immediately prior to study enrollment.
* Hepatic insufficiency (elevated transaminases > 1.5 times the upper limit of normal) or renal insufficiency (plasma creatinine > 2mg/dl).
* Known or suspected history of alcohol or illicit drug abuse.
* Pregnant or breast-feeding.
* Surgical plan for infratentorial (suboccipital) craniotomy.
* Plan for neurophysiologic monitoring that precludes the use of neuromuscular blockade.
* Inability to communicate due to a language barrier, impaired consciousness, cognitive defect or intellectual disability.
* Uncontrolled Hypertension

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05-02 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2016-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A. Artime, MD, Principal Investigator — University of Texas Health Sciences Center at Houston; Sam D. Gumbert, MD, Principal Investigator — University of Texas Health Sciences Center at Houston
Locations (1):
- Memorial Hermann Hospital - Texas Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Artime CA, Aijazi H, Zhang H, Syed T, Cai C, Gumbert SD, Ferrario L, Normand KC, Williams GW, Hagberg CA. Scheduled Intravenous Acetaminophen Improves Patient Satisfaction With Postcraniotomy Pain Management: A Prospective, Randomized, Placebo-controlled, Double-blind Study. J Neurosurg Anesthesiol. 2018 Jul;30(3):231-236. doi: 10.1097/ANA.0000000000000461. PMID 29117012

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous Acetaminophen | Placebo
Started | 50 | 50
Completed | 45 | 41
Not Completed | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Acetaminophen | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (16.3) | 51.5 (14.4) | 50.75 (15.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 31 | 55
  Male | 26 | 19 | 45

OUTCOME MEASURES:

1. Primary Outcome: Post-Operative Opioid Requirement
Description: Opioid Consumption will be monitored in the first 24 post-operative hours. All non-opioid analgesics are disallowed. Total opioid consumption was calculated based on morphine equivalents (MEs), where 1 mg of IV morphine was equivalent to 1 ME, and 1 mg IV hydromorphone was calculated as 7 MEs.
Time Frame: 24 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: Morphine Equivalents
Arm/Group | Intravenous Acetaminophen | Placebo
Number analyzed (Participants) | 45 | 41
Morphine Equivalents | 11.0 [2 to 21] | 10.1 [1 to 16.7]

2. Secondary Outcome: Post-Operative Pain
Description: Patients will be assessed for pain using a Visual Analogue Scale (VAS) Scale at set time points after surgery (0,1,2,4,8,12,16,20,24 hours post-operatively). The Visual Analogue Scale (VAS) scale was measured on a scale of 0 - 10 (0 = no pain, 1-3 = mild, 4-6 = moderate, 7-10 = severe). Higher values on the VAS represent a worse outcome. The two rows below report: 1. the average VAS score for the least amount of pain reported per group and 2. the average VAS score of the worst amount of pain reported per group.
Time Frame: 24 Hours Post-Operatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Acetaminophen | Placebo
Number analyzed (Participants) | 45 | 41
units on a scale
  Least amount of pain reported | 1.4 (1.8) | 2.6 (2.7)
  Worst amount of pain reported | 6.3 (2.5) | 6.4 (3.2)

3. Secondary Outcome: Post-Operative Side Effects
Description: Patients will be monitored for 24 hours post-operatively to detect the incidence of any drug or opioid-related side effects. These side effects were not considered to be adverse events.
Time Frame: 24 Hours Post-Operatively
Population: The # analyzed does not match the # who completed or the overall # analyzed because data on all side effects was not collected for all participants who completed, either due to lack of collection of data by research/nursing staff (for emesis) or due to lack of reporting by participants on a questionnaire(for itching, dizziness, and drowsiness).
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Acetaminophen | Placebo
Number analyzed (Participants) | 45 | 40
Participants
  Emesis | 23 | 20
  Itching: number analyzed (Participants) | 42 | 37
  Itching | 8 | 5
  Dizziness: number analyzed (Participants) | 42 | 37
  Dizziness | 14 | 14
  Drowsiness: number analyzed (Participants) | 42 | 37
  Drowsiness | 24 | 19

4. Secondary Outcome: Time to Extubation at Emergence From Anesthesia
Time Frame: Time from of discontinuation of anesthetic to time of extubation, an average of 7 minutes
Population: The number analyzed is greater than the number completed because this data was collected for more patients than completed the study, and all data that was collected is reported here.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Intravenous Acetaminophen | Placebo
Number analyzed (Participants) | 48 | 45
minutes | 6 [3 to 13] | 8 [5 to 12]

5. Secondary Outcome: Time for Patient to Meet Post-anesthesia Care Unit (PACU) Discharge Criteria
Time Frame: From time of entry to PACU to time to meet PACU discharge criteria, an average of 12 minutes
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intravenous Acetaminophen | Placebo
Number analyzed (Participants) | 46 | 43
minutes | 11.4 (7.2) | 13.5 (8.4)

ADVERSE EVENTS:
Arm/Group | Intravenous Acetaminophen | Placebo
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 1/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Acetaminophen (N=50) | Placebo (N=50)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Not powered to detect differences in pain score. Patients were not given a patient-controlled analgesia device; rather, administration of morphine was dependent on nurse administration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No